CLINICAL TRIAL: NCT02334228
Title: Promoting Health and Functioning in Persons With SMI
Brief Title: Evaluation of the In SHAPE Fitness Intervention for Adults With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Concord InSHAPE
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder; Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders; Depressive Disorder, Major | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In SHAPE Lifestyles (Experimental): In SHAPE Lifestyle is a health promotion intervention consisting of a fitness club membership and a health promotion coach with basic certification as a fitness trainer, instruction on principles of healthy eating and nutrition, and training in tailoring individual wellness plans to the needs of persons with serious mental illness.
  Interventions: Behavioral: In SHAPE Lifestyles
- Health Club Membership and Education (Active Comparator): Fitness club membership with education in using the exercise equipment.
  Interventions: Behavioral: Health Club Membership and Education

INTERVENTIONS:
Behavioral: In SHAPE Lifestyles — In SHAPE Lifestyles is a health promotion intervention consisting of a fitness club membership and a health promotion coach with basic certification as a fitness trainer, instruction on principles of healthy eating and nutrition, and training in tailoring individual wellness plans to the needs of persons with serious mental illness.
  Arms: In SHAPE Lifestyles
Behavioral: Health Club Membership and Education — Fitness club membership with education in using the exercise equipment.
  Arms: Health Club Membership and Education

SUMMARY:
Few studies targeting obesity in serious mental illness have reported clinically significant risk reduction, and non have been replicated in community settings or demonstrated sustained outcomes after intervention withdrawal. The researchers sought to replicate positive health outcomes demonstrated in a previous randomized effectiveness study of the In SHAPE program across urban community mental health organizations serving an ethnically diverse population.

DETAILED DESCRIPTION:
In this randomized, controlled study, 133 adults age 21 and older with serious mental illness (SMI) and poor physical fitness (BMI>25, or <10 minutes of exercise 2x over the past month) were randomized to either: a) In SHAPE Lifestyles (ISL) intervention or b) Health Club Membership and Education (HCME): consisting of a YMCA membership, educational materials on exercise and healthy diet, and an on-site introduction to the health club. The following three specific aims were addressed: 1) To compare ISL and HCME with respect to: a) participation in regular exercise and dietary change; (b) participation in preventive health care; and (c) improved fitness and health; (2) to compare ISL and HCME with respect to: (a) indicators of mental health and (b) personal self-efficacy; and (3) to explore differences in ISL and HCME with respect to (a) selected physical, metabolic, dietary, and community functioning secondary outcomes; and (b) the relationship of demographic variables and readiness to change to outcomes. ISL participants received a 6-month intensive program of one-to-one health mentoring, followed by a 3-month period of transitioning to self-directed individual and group programming, with assessments conducted at baseline, 3, 6, 9, and 12 months. If found to be effective, ISL will provide a practical approach to improving health, independent functioning, and longevity in disabled persons with SMI.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Serious mental illness defined by an axis I diagnosis of major depression, bipolar disorder, schizoaffective disorder, or schizophrenia
* Persistent impairment in multiple areas of functioning (e.g., work, school, self-care)
* Body mass index (BMI) greater than 25
* Able and willing to provide informed consent
* On stable pharmacological treatment (same psychiatric medications over prior 2 months)

Exclusion Criteria:

* Residing in a nursing home of other institution
* Diagnosis of dementia or significant cognitive impairment (MMSE<24)
* Unable to walk one city block
* Pregnant or planning to become pregnant within the next 18 months
* Unable to speak English
* Terminal illness with life expectancy <1 year
* Current diagnosis of an active substance dependence disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in Exercise Capacity | Baseline, 3-, 6-, 9-, and 12-months
  Change in fitness as measured by the 6-minute walk test.

SECONDARY OUTCOMES:
Body Mass Index | Baseline, 3-, 6-, 9-, and 12-months
Change in Weight | Baseline, 3-, 6-, 9-, and 12-months
  Change in weight over time was measured at baseline, 3-, 6-, 9-, and 12-months. Measures were weight (lbs).
Change in Triglycerides and Cholesterol | Baseline, 3-, 6-, 9-, and 12-months
  Change in triglycerides and cholesterol measured with the CardioChek PA Analyzer: Fasting blood glucose and lipids.
Change in Health Status | Baseline, 3-, 6-, 9-, and 12-months
  Change in health status was measured by the SF-12: Medical Outcomes Study Short Form -12
Change in Community Functioning | Baseline, 9-, and 12-months
  Change in community functioning was measured by the ILSS: Independent Living Skills Scale
Change in Physical Measurements (Fitness) | Baseline, 3-, 6-, 9-, and 12-months
  Change is physical measurements was determined by measuring waist circumference and resting pulse
Change in Psychological State | Baseline, 3-, 6-, 9-, and 12-months
  Change in psychological state was measured using the CESD: Cntr Epid Studies Dep; SANS: Scale Assess Neg Sx; R-SES: Revised Self-efficacy Scale
Change in Participation in Exercise | Baseline, 3-, 6-, 9-, and 12-months
  Change in participation in exercise was determined by measuring weekly exercise at 3-, 6-, 9-, and 12-months using a physical activity log; weekly health club attendance at 3-, 6-, 9-, and 12-months based on frequency of YMCA visits; total physical activity at baseline, 3-, 6-, 9-, and 12-months based on the YPAS: Yale Physical Activity Scale.
Change in Diet Behaviors | Baseline, 3-, 6-, 9-, and 12-months
  Change in diet behaviors was measured based on the WLB-SOC: Weight Loss Behavior State of Change Scale.
Change in Preventative Health Care | Baseline and 12-months
  Change in preventative health care was based on the PHC: Preventative Healthcare Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bartels, MD,MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Riverbend Community Mental Health, Concord, New Hampshire, United States